CLINICAL TRIAL: NCT01375764
Title: A Randomized, Multicenter Study to Evaluate Tolerability and Efficacy of AMG 145 on LDL-C, Compared With Ezetimibe, in Hypercholesterolemic Subjects Unable to Tolerate an Effective Dose of a HMG-CoA Reductase Inhibitor
Brief Title: Goal Achievement After Utilizing an Anti-PCSK9 Antibody in Statin Intolerant Subjects
Acronym: GAUSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20090159
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Hyperlipidemia
Keywords: Proprotein convertase subtilisin/kexin type 9 (PCSK9); Cholesterol; High Cholesterol; Raised Cholesterol; Elevated Cholesterol; Statin intolerant; Hypercholesterolemia
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia, Autosomal Dominant, 3; Hypercholesterolemia | interventions — evolocumab; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Ezetimibe (Active Comparator): Participants received placebo subcutaneous injection once every 4 weeks and 10 mg ezetimibe orally once a day for 12 weeks.
  Interventions: Drug: Ezetimibe; Other: Placebo to Evolocumab
- Evolocumab + Ezetimibe (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once every 4 weeks and 10 mg ezetimibe orally once a day for 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Ezetimibe
- Evolocumab 280 mg (Experimental): Participants received 280 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 350 mg (Experimental): Participants received 350 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 420 mg (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: Evolocumab + Ezetimibe; Evolocumab 280 mg; Evolocumab 350 mg; Evolocumab 420 mg
Drug: Ezetimibe — Administered orally once a day
  Other Names: Zetia
  Arms: Evolocumab + Ezetimibe; Ezetimibe
Other: Placebo to Evolocumab — Administered by subcutaneous injection
  Arms: Ezetimibe

SUMMARY:
The primary objective was to evaluate the effect of 12 weeks of subcutaneous evolocumab (AMG 145), compared with ezetimibe, on percent change from baseline in low-density lipoprotein cholesterol (LDL-C) in patients with hypercholesterolemia unable to tolerate an effective dose of a statin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 to ≤ 75 years of age
* On a statin or a low dose statin with stable dose for at least 4 weeks
* Lipid lowering therapy has been stable prior to enrollment
* Fasting triglycerides must be < 400 mg/dL.
* Subject not at LDL-C goal

Exclusion Criteria:

* New York Heart Association (NYHA) III or IV heart failure or known left ventricular ejection fraction < 30%
* Uncontrolled cardiac arrhythmia
* Myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or stroke within 3 months prior to randomization
* Type 1 diabetes or newly diagnosed type 2 diabetes (HbA1c > 8.5%)
* Uncontrolled hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-07-28 (Actual); Primary Completion 2012-05-08 (Actual); Study Completion 2012-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (40):
- United States (15):
  - Research Site, Anaheim, California
  - Research Site, Mission Viejo, California
  - Research Site, Westlake Village, California
  - Research Site, Atlanta, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Auburn, Maine
  - Research Site, Chevy Chase, Maryland
  - Research Site, Butte, Montana
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Bristol, Tennessee
- Australia (4):
  - Research Site, Camperdown, New South Wales
  - Research Site, Sydney, New South Wales
  - Research Site, Melbourne, Victoria
  - Research Site, Perth, Western Australia
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Uccle
- Canada (3):
  - Research Site, Saint Johnâ€™s, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Lachine, Quebec
- Denmark (2):
  - Research Site, Ballerup Municipality
  - Research Site, Vejle
- Finland (2):
  - Research Site, Helsinki
  - Research Site, OYS
- Spain (8):
  - Research Site, Zaragoza, Aragon
  - Research Site, Zaragoza, AragÃ³n
  - Research Site, Barcelona, Catalonia
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, Reus, Catalonia
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, L'Hospitalet de Llobregat, CataluÃ±a
  - Research Site, Reus, CataluÃ±a
- Sweden (4):
  - Research Site, GÃ¶teborg
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Stockholm

REFERENCES:
- [Background] Sullivan D, Olsson AG, Scott R, Kim JB, Xue A, Gebski V, Wasserman SM, Stein EA. Effect of a monoclonal antibody to PCSK9 on low-density lipoprotein cholesterol levels in statin-intolerant patients: the GAUSS randomized trial. JAMA. 2012 Dec 19;308(23):2497-506. doi: 10.1001/jama.2012.25790. PMID 23128163
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled adults aged 18 to 75 years with hypercholesterolemia who were statin intolerant and with low-density lipoprotein cholesterol (LDL-C) levels above risk-based goals recommended by the National Cholesterol Education Program.
  The first patient enrolled on 28 July 2011; last patient enrolled 14 February 2012.
Pre-assignment Details: Randomization was stratified by screening LDL-C level (< 130 mg/dL [3.4 mmol/L] or ≥ 130 mg/dL) and statin use at baseline (yes or no).
Period: Overall Study
Arm/Group | Ezetimibe | Evolocumab + Ezetimibe | Evolocumab 280 mg | Evolocumab 350 mg | Evolocumab 420 mg
Started | 33 | 31 | 32 | 32 | 32
Received Treatment | 32 | 30 | 32 | 31 | 32
Completed | 31 | 30 | 32 | 31 | 31
Not Completed | 2 | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (all randomized participants who received at least 1 dose of investigational product).
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe | Evolocumab + Ezetimibe | Evolocumab 280 mg | Evolocumab 350 mg | Evolocumab 420 mg | Total
Number analyzed (Participants) | 32 | 30 | 32 | 31 | 32 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (6.6) | 62.0 (7.2) | 62.2 (10.1) | 62.3 (9.1) | 60.0 (8.6) | 61.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 18 | 21 | 20 | 100
  Male | 14 | 7 | 14 | 10 | 12 | 57
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 5 | 1 | 0 | 0 | 8
  Black or African American | 2 | 1 | 2 | 2 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  White | 28 | 24 | 28 | 29 | 30 | 139
  Other | 0 | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 30 | 30 | 32 | 31 | 32 | 155
Stratification Factor: LDL-C Level [Number; unit: participants]
  < 130 mg/dL | 2 | 1 | 2 | 2 | 2 | 9
  ≥ 130 mg/dL | 30 | 29 | 30 | 29 | 30 | 148
Stratification Factor: Baseline Use of Statin [Number; unit: participants]
  No | 26 | 26 | 27 | 27 | 27 | 133
  Yes | 6 | 4 | 5 | 4 | 5 | 24
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] | 182.9 (36.4) | 194.4 (60.1) | 194.8 (48.1) | 190.3 (47.8) | 203.5 (60.3) | 193.2 (51.0)
Non-High-Density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 213.7 (40.4) | 219.8 (60.5) | 225.5 (53.3) | 222.9 (55.8) | 240.6 (63.9) | 224.6 (55.3)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] | 138.0 (21.7) | 138.8 (33.1) | 143.0 (30.6) | 144.9 (33.9) | 150.8 (34.1) | 143.2 (30.9)
Total Cholesterol/HDL-C Ratio [Mean (Standard Deviation); unit: ratio] | 4.907 (1.553) | 5.093 (2.416) | 5.287 (1.816) | 5.444 (2.308) | 6.438 (2.834) | 5.438 (2.265)
Apolipoprotein B/Apolipoprotein A-1 Ratio [Mean (Standard Deviation); unit: ratio] | 0.841 (0.230) | 0.882 (0.332) | 0.906 (0.265) | 0.916 (0.332) | 1.055 (0.388) | 0.921 (0.319)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: LDL-C was measured using ultracentrifugation. Least squares (LS) means are based off an analysis of covariance (ANCOVA) model which includes treatment group (3 evolocumab alone dose groups and the ezetimibe group) and stratification factors as covariates.
Time Frame: Baseline and Week 12
Population: Full analysis set; Missing ultracentrifugation (UC) LDL-C at Week 12 was imputed using last observation carried forward (LOCF) and calculated LDL-C.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab 280 mg | Evolocumab 350 mg | Evolocumab 420 mg
Number analyzed (Participants) | 32 | 32 | 31 | 32
percent change | -14.76 (3.94) | -40.77 (3.96) | -42.58 (4.01) | -50.70 (3.98)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab 420 mg; The null hypothesis was that there was no mean difference in the percent change from Baseline at Week 12 in LDL-C between evolocumab and ezetimibe, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group (3 evolocumab alone dose groups and the ezetimibe group) and the stratification factors; LS Mean Treatment Difference = -35.94, 95% CI 2-sided [-44.08 to -27.80], Standard Error of Mean 4.11 — Ezetimibe is the reference
Statistical Analysis 2: Comparison: Ezetimibe vs Evolocumab 350 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.82, 95% CI 2-sided [-35.97 to -19.67], Standard Error of Mean 4.12 — Ezetimibe is the reference
Statistical Analysis 3: Comparison: Ezetimibe vs Evolocumab 280 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Tretament Difference = -26.01, 95% CI 2-sided [-34.08 to -17.93], Standard Error of Mean 4.08 — Ezetimibe is the reference

2. Primary Outcome: Percent Change From Baseline in LDL-C at Week 12: Ezetimibe Alone Versus Evolocumab + Ezetimibe
Description: LDL-C was measured using ultracentrifugation. LS means are based off an ANCOVA model which includes treatment group (evolocumab + ezetimibe and ezetimibe alone) and stratification factors as covariates.
Time Frame: Baseline and Week 12
Population: Full analysis set; Missing UC LDL-C at Week 12 was imputed using LOCF and calculated LDL-C.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab + Ezetimibe
Number analyzed (Participants) | 32 | 30
percent change | -15.70 (3.98) | -62.98 (4.22)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab + Ezetimibe; The null hypothesis was that there was no mean difference in the percent change from Baseline at Week 12 in LDL-C between evolocumab + ezetimibe and ezetimibe alone, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group (evolocumab + ezetimibe and ezetimibe alone) and the stratification factors; LS Mean Treatment Difference = -47.29, 95% CI 2-sided [-53.73 to -40.84], Standard Error of Mean 3.22 — Ezetimibe is the reference

3. Secondary Outcome: Change From Baseline in LDL-C at Week 12
Description: LDL-C was measured using ultracentrifugation. LS means are based off an ANCOVA model which includes treatment group (3 evolocumab alone dose groups and the ezetimibe group) and stratification factors as covariates.
Time Frame: Baseline and Week 12
Population: Full analysis set; Missing UC LDL-C at Week 12 was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Ezetimibe | Evolocumab 280 mg | Evolocumab 350 mg | Evolocumab 420 mg
Number analyzed (Participants) | 32 | 32 | 31 | 32
mg/dL | -14.2 (8.9) | -66.8 (8.9) | -69.7 (9.1) | -90.8 (9.0)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab 420 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -76.6, 95% CI 2-sided [-94.9 to -58.3], Standard Error of Mean 9.2 — Ezetimibe is the reference
Statistical Analysis 2: Comparison: Ezetimibe vs Evolocumab 350 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -55.5, 95% CI 2-sided [-74.0 to -37.1], Standard Error of Mean 9.3 — Ezetimibe is the reference
Statistical Analysis 3: Comparison: Ezetimibe vs Evolocumab 280 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -52.6, 95% CI 2-sided [-70.8 to -34.5], Standard Error of Mean 9.2 — Ezetimibe is the reference

4. Secondary Outcome: Change From Baseline in LDL-C at Week 12: Ezetimibe Alone Versus Evolocumab + Ezetimibe
Description: LDL-C was measured using ultracentrifugation. LS means are based off an ANCOVA model which includes treatment group (evoloumab + ezetimibe and ezetimibe alone) and stratification factors as covariates.
Time Frame: Baseline and Week 12
Population: Full analysis set; Missing UC LDL-C at Week 12 was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Ezetimibe | Evolocumab + Ezetimibe
Number analyzed (Participants) | 32 | 30
mg/dL | -17.9 (10.4) | -109.8 (11.0)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab + Ezetimibe; Test type: Superiority or Other; p < 0001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group (evolocumab + ezetimibe and ezetimibe alone) and the stratification factors; LS Mean Treatment Difference = -91.9, 95% CI 2-sided [-108.7 to -75.0], Standard Error of Mean 8.4 — Ezetimibe is the reference

5. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12
Description: LS means are based off an ANCOVA model which includes treatment group (3 evolocumab alone dose groups and the ezetimibe group) and stratification factors as covariates.
Time Frame: Baseline and Week 12
Population: Full analysis set; missing non-HDL-C at Week 12 was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab 280 mg | Evolocumab 350 mg | Evolocumab 420 mg
Number analyzed (Participants) | 32 | 32 | 31 | 32
percent change | -14.97 (3.54) | -39.83 (3.56) | -41.63 (3.61) | -48.58 (3.58)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab 420 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -33.60, 95% CI 2-sided [-40.93 to -26.28], Standard Error of Mean 3.70 — Ezetimibe is the reference
Statistical Analysis 2: Comparison: Ezetimibe vs Evolocumab 350 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -26.66, 95% CI 2-sided [-33.99 to -19.32], Standard Error of Mean 3.70 — Ezetimibe is the reference
Statistical Analysis 3: Comparison: Ezetimibe vs Evolocumab 280 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -24.86, 95% CI 2-sided [-32.13 to -17.59], Standard Error of Mean 3.67 — Ezetimibe is the reference

6. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12: Ezetimibe Alone Versus Evolocumab + Ezetimibe
Description: LS means are based off an ANCOVA model which includes treatment group (evolocumab + ezetimibe and ezetimibe alone) and stratification factors as covariates.
Time Frame: Baseline and Week 12
Population: Full analysis set; missing non-HDL-C at Week 12 was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab + Ezetimibe
Number analyzed (Participants) | 32 | 30
percent change | -14.83 (3.59) | -59.82 (3.81)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab + Ezetimibe; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group (evolocumab + ezetimibe and ezetimibe alone) and the stratification factors; LS Mean Treatment Difference = -45.00, 95% CI 2-sided [-50.81 to -39.18], Standard Error of Mean 2.90 — Ezetimibe is the reference

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 12
Description: as for outcome 5
Time Frame: Baseline and Week 12
Population: Full analysis set; missing Apolipoprotein B at Week 12 was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab 280 mg | Evolocumab 350 mg | Evolocumab 420 mg
Number analyzed (Participants) | 32 | 32 | 31 | 32
percent change | -12.20 (3.37) | -33.58 (3.39) | -34.33 (3.43) | -42.07 (3.40)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab 420 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Teatment Difference = -29.88, 95% CI 2-sided [-36.84 to -22.92], Standard Error of Mean 3.52 — Ezetimibe is the reference
Statistical Analysis 2: Comparison: Ezetimibe vs Evolocumab 350 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -22.13, 95% CI 2-sided [-29.10 to -15.16], Standard Error of Mean 3.52 — Ezetimibe is the reference
Statistical Analysis 3: Comparison: Ezetimibe vs Evolocumab 280 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a signficance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -21.38, 95% CI 2-sided [-28.29 to -14.48], Standard Error of Mean 3.49 — Ezetimibe is the reference

8. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 12: Ezetimibe Alone Versus Evolocumab + Ezetimibe
Description: LS means are based off an ANCOVA model which includes treatment group (evoloumab + ezetimibe and ezetimibe) and stratification factors as covariates.
Time Frame: Baseline and Week 12
Population: Full analysis set; missing Apolipoprotein B at Week 12 was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab + Ezetimibe
Number analyzed (Participants) | 32 | 30
percent change | -10.84 (3.45) | -49.06 (3.66)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab + Ezetimibe; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group (evolocumab + ezetimibe and ezetimibe alone) and the stratification factors; LS Mean Treatment Difference = -38.23, 95% CI 2-sided [-43.81 to -32.64], Standard Error of Mean 2.79 — Ezetimibe is the reference

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol/HDL-C Ratio at Week 12
Description: as for outcome 5
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data at Week 12 were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab 280 mg | Evolocumab 350 mg | Evolocumab 420 mg
Number analyzed (Participants) | 32 | 32 | 31 | 32
percent change | -9.61 (3.20) | -31.97 (3.22) | -33.52 (3.26) | -40.56 (3.23)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab 420 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -30.95, 95% CI 2-sided [-37.56 to -24.34], Standard Error of Mean 3.34 — Ezetimibe is the reference
Statistical Analysis 2: Comparison: Ezetimibe vs Evolocumab 350 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -23.91, 95% CI 2-sided [-30.53 to -17.29], Standard Error of Mean 3.34 — Ezetimibe is the reference
Statistical Analysis 3: Comparison: Ezetimibe vs Evolocumab 280 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -22.36, 95% CI 2-sided [-28.92 to -15.80], Standard Error of Mean 3.31 — Ezetimibe is the reference

10. Secondary Outcome: Percent Change From Baseline in Total Cholesterol/HDL-C Ratio at Week 12: Ezetimibe Alone Versus Evolocumab + Ezetimibe
Description: LS means are based off an ANCOVA model which includes treatment group (evoloumab + ezetimibe and ezetimibe alone) and stratification factors as covariates.
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data at Week 12 were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab + Ezetimibe
Number analyzed (Participants) | 32 | 30
percent change | -11.52 (3.61) | -49.44 (3.83)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab + Ezetimibe; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group (evolocumab + ezetimibe and ezetimibe alone) and the stratification factors; LS Mean Treatment Difference = -37.92, 95% CI 2-sided [-43.77 to -32.07], Standard Error of Mean 2.92 — Ezetimibe is the reference

11. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at Week 12
Description: as for outcome 5
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data at Week 12 were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab 280 mg | Evolocumab 350 mg | Evolocumab 420 mg
Number analyzed (Participants) | 32 | 32 | 31 | 32
percent change | -11.36 (3.16) | -36.46 (3.18) | -38.17 (3.22) | -45.41 (3.19)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab 420 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -34.05, 95% CI 2-sided [-40.57 to -27.52], Standard Error of Mean 3.30 — Ezetimibe is the reference
Statistical Analysis 2: Comparison: Ezetimibe vs Evolocumab 350 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -26.81, 95% CI 2-sided [-33.35 to -20.27], Standard Error of Mean 3.30 — Ezetimibe is the reference
Statistical Analysis 3: Comparison: Ezetimibe vs Evolocumab 280 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -25.10, 95% CI 2-sided [-31.57 to -18.62], Standard Error of Mean 3.27 — Ezetimibe is the reference

12. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at Week 12: Ezetimibe Alone Versus Evolocumab + Ezetimibe
Description: as for outcome 10
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data at Week 12 were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe | Evolocumab + Ezetimibe
Number analyzed (Participants) | 32 | 30
percent change | -10.74 (3.55) | -51.99 (3.76)
Statistical Analysis 1: Comparison: Ezetimibe vs Evolocumab + Ezetimibe; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group (evolocumab + ezetimibe and ezetimibe alone) and the stratification factors; LS Mean Treatment Difference = -41.25, 95% CI 2-sided [-46.99 to -35.50], Standard Error of Mean 2.87 — Ezetimibe is the reference

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Ezetimibe | Evolocumab 280 mg | Evolocumab 350 mg | Evolocumab 420 mg | Evolocumab + Ezetimibe
Serious Adverse Events (participants affected / at risk) | 0/32 | 2/32 | 1/31 | 1/32 | 0/30
Other Adverse Events (participants affected / at risk) | 16/32 | 19/32 | 10/31 | 12/32 | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ezetimibe (N=32) | Evolocumab 280 mg (N=32) | Evolocumab 350 mg (N=31) | Evolocumab 420 mg (N=32) | Evolocumab + Ezetimibe (N=30)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ezetimibe (N=32) | Evolocumab 280 mg (N=32) | Evolocumab 350 mg (N=31) | Evolocumab 420 mg (N=32) | Evolocumab + Ezetimibe (N=30)
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 0
Fatigue (General disorders) | 2 | 4 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Influenza (Infections and infestations) | 2 | 0 | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 5 | 2 | 2 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 2
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 1 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 3
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.